CLINICAL TRIAL: NCT00034840
Title: A Prospective, Randomized, Double-Blind, Forced Titration Trial to Compare the Efficacy of MICARDIS® (Telmisartan 80 mg p.o. Once Daily) and Diovan® (Valsartan 160 mg p.o. Once Daily) Using Ambulatory Blood Pressure Monitoring (ABPM) in Patients With Mild to Moderate Hypertension After Missing One Dose
Brief Title: Telmisartan vs. Valsartan in Patients With Mild to Moderate Hypertension Following a Missed Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: GlaxoSmithKline (Industry); Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.327
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
Keywords: hypertension; telmisartan; valsartan; boehringer
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Valsartan

INTERVENTIONS:
Drug: telmisartan, valsartan

SUMMARY:
The primary objectives are to demonstrate that MICARDIS® (telmisartan) is statistically superior to Diovan® (valsartan) in reducing diastolic blood pressure (DBP) following a missed dose at the end of a 6 to 8-week treatment period as measured by the 24-hour ABPM mean and to demonstrate that MICARDIS® is statistically superior to Diovan® in reducing DBP during the last 6-hours of the 24-hour dosing interval as measured by ABPM following a dose of active study medication at the end of a 6 to 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Mild-to-moderate hypertension defined as a baseline mean seated DBP of greater than or equal to 95 mm Hg and less than or equal to 109 mm Hg and a baseline 24-hour ABPM mean DBP of greater than or equal to 85 mm Hg.

Exclusion Criteria:

1. Pre-menopausal women (last menstruation = 1 year prior to signing informed consent) who:

   * Are not surgically sterile.
   * Are nursing.
   * Are of child-bearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control include IUD, oral, implantable or injectable contraceptives. No exceptions will be made.
2. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 A.M.
3. Mean sitting SBP =180 mm Hg or mean sitting DBP =110 mm Hg during any visit of the placebo run-in period.
4. Known or suspected secondary hypertension (i.e., pheochromocytoma).
5. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT (ALT) or SGOT (AST) > 2 times the upper limit of normal range.
   * Serum creatinine > 2.3 mg/dL (or > 203 µmol/l).
6. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney.
7. Clinically relevant sodium depletion, hypokalaemia or hyperkalaemia.
8. Uncorrected volume depletion.
9. Primary aldosteronism.
10. Hereditary fructose intolerance.
11. Biliary obstructive disorders.
12. Congestive heart failure (NYHA functional class CHF III-IV).
13. Unstable angina within the past three months prior to signing the informed consent form.
14. Stroke within the past six months prior to signing the informed consent form.
15. Myocardial infarction or cardiac surgery within the past three months prior to signing the informed consent form.
16. PTCA (percutaneous transluminal coronary revascularization) within the past three months prior to signing the informed consent form.
17. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator.
18. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve.
19. Patients with insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C =10%.
20. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists.
21. History of drug or alcohol dependency within 6 months prior to signing the informed consent form.
22. Chronic administration of any medications known to affect blood pressure, except medication allowed by the protocol.
23. Any investigational therapy within one month of signing the informed consent form.
24. Known hypersensitivity to any component of the formulations.
25. Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication.
26. Inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490
Dates: Start 2001-10; Primary Completion 2002-08 (Actual); Study Completion 2002-08

PRIMARY OUTCOMES:
Change in the 24-hour mean diastolic blood pressure (DBP), as measured by ABPM after a missed dose | after 6 to 8 weeks
Change in the mean DBP during the last 6 hours of the 24-hour dosing interval, as measured by ABPM after an active dose of study medication | after 6 to 8 weeks

SECONDARY OUTCOMES:
Change in 24-hour ABPM mean systolic blood pressure (SBP) after a missed dose | after 6 to 8 weeks
Change in the last 6 hour ABPM mean SBP measured after a dose of active treatment | after 6 to 8 weeks
Changes in ABPM mean DBP and SBP during other periods of the 24-hour dosing interval after an active dose | 8 weeks
Changes in ABPM mean DBP and SBP during other periods of the 24-hour dosing interval after a missed dose | 8 weeks
Changes in in-clinic mean seated trough DBP and SBP as measured by manual cuff sphygmomanometer after a missed dose | 8 weeks
Changes in in-clinic mean seated trough DBP and SBP as measured by manual cuff sphygmomanometer after an active dose | 8 weeks
Responder rates based on ABPM | after 6 to 8 weeks
Responder rates based on in-clinic trough cuff blood pressures | after 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (35):
- United States (16):
  - Memorial Research Medical Clinic, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Orange County Research Center, Orange, California
  - University of Conn. Health Services Center, Hypertension and Vascular Disease, Farmington, Connecticut
  - Alan Graff, Fort Lauderdale, Florida
  - Greater Ft. Lauderdale Heart Group Research, Fort Lauderdale, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - So. Clinical Research and Management, Inc., Augusta, Georgia
  - Rush Presbyterian/St. Luke's Medical Center, Chicago, Illinois
  - University of Maryland/Nephrology Clinical Research Unit, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Oklahoma Cardiovascular and Hypertension Center, Oklahoma City, Oklahoma
  - Michael A. Azorr, M.D., Portland, Oregon
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Trinity Hypertension Research Institute/Punzi Medical Center, Carrollton, Texas
  - UW Health/Physicians Plus Center for Clinical Trials, Madison, Wisconsin
- Canada (19):
  - Heart Health Institute, Calgary, Alberta
  - Dr. Dennis O'Keefe, Mount Pearl, Newfoundland and Labrador
  - Dr. William Booth, Antigonish, Nova Scotia
  - MSHJ Research Assoc., Halifax, Nova Scotia
  - Dr. Joseph Berlingieri, Burlington, Ontario
  - Dr. William Mahoney, Corunna, Ontario
  - BBM Clinical Research Ltd., Courtice, Ontario
  - Dr. Richard Tytus, Hamilton, Ontario
  - Total Concept Health Care, Kitchener, Ontario
  - Centre for Activity and Aging, London, Ontario
  - Dr. Martyn Chilvers, Sarnia, Ontario
  - Sunnybrook & Women's College Health Centre, Toronto, Ontario
  - Theradev Clinical Research, Inc., Granby, Quebec
  - Invascor, Longueuil, Longueuil, Quebec
  - Hotel Dieu de St-Jerome, Saint-Jérôme, Quebec
  - Centre de Cardiologie, Saint-Lambert, Quebec
  - Centre Hospital Quebec - PAC CHUL Unite de Recherche, Sainte-Foy, Quebec
  - Q&T Research, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan